CLINICAL TRIAL: NCT00453427
Title: Alemtuzumab and CHOP Chemotherapy for Aggressive Histological Peripheral T-Cell Lymphomas: A Multi-centre Phase I and II Study
Brief Title: Alemtuzumab and CHOP Chemotherapy for Aggressive Histological Peripheral T-Cell Lymphomas
Acronym: ACCAPELA
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ontario Clinical Oncology Group (OCOG) (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTA-Control-103662
Record Dates: First submitted 2007-03-27; First posted 2007-03-29 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Peripheral T-cell Lymphomas
Keywords: PTL NOS; AILD; NHL; CHOP
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — Alemtuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Alemtuzumab (Campath-1H) — The investigational drug is alemtuzumab (Campath-1H). It is a recombinant humanized monoclonal antibody directed against the CD52 antigen on most (> 95%) normal lymphocytes and T-cell and B-cell lymphomas. Alemtuzumab binds to the CD52 antigen on the cell surface, activating antibody-dependent cellular cytotoxicity, complement binding, apoptosis, cellular opsonization, and anti-tumour T-cell activity.

SUMMARY:
The primary objectives of this study are to:

1. establish the safety and dose limiting toxicities of combining alemtuzumab with CHOP chemotherapy for patients with newly diagnosed aggressive T-cell lymphomas; and
2. to measure the pharmacokinetics of alemtuzumab used in different subcutaneous doses and schedules.

This will then determine the dose with the highest achievable drug levels with acceptable toxicities worthy of further investigation.

The secondary objectives are to:

1. establish the efficacy of combination alemtuzumab with CHOP chemotherapy; and
2. to measure the effects of combination alemtuzumab with CHOP chemotherapy on T-cell reconstitution and cytomegalovirus (CMV) reactivation.

DETAILED DESCRIPTION:
Aggressive peripheral T-cell lymphomas account for 10 - 15% of all Non-Hodgkin's Lymphoma (NHL) and present with more adverse prognostic features than aggressive histology B-cell NHL . Correspondingly, they have an overall poorer prognosis than B-cell lymphomas, achieving lower complete response rates, freedom from progression and overall survival with conventional anthracycline-based CHOP (cyclophosphamide, doxorubicin, vincristine and prednisone) chemotherapy. Fewer than 30% of patients are cured with therapy. New treatments that replicate the improved survivals with chemo-immunotherapy for B-cell lymphomas are needed. Alemtuzumab is a humanized murine antibody that binds to a ubiquitous lymphoid marker CD52 and is efficacious (as monotherapy) in related lymphoproliferative diseases. Combining alemtuzumab with CHOP chemotherapy may improve the response rates and outcomes of patients with this sub-type of NHL. The combination must be first tested in a dose escalation fashion to establish the dosage of the doublet because of the potential for overlapping or exaggerated toxicities.

This prospective, multi-center, open label Phase I-II study will enroll 22-84 patients with newly diagnosed previously untreated aggressive histology peripheral T-cell lymphomas. In the Phase I component, patients will be sequentially enrolled in cohorts of three patients and treated with increasing doses of alemtuzumab administered in combination with standard CHOP chemotherapy. When the maximal tolerated dose is determined, this dose and schedule will then be tested in up to 46 patients using a Simon two stage Phase II design.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years of age or older at time of enrollment,
* Histologically proven and centrally reviewed CD52+ T-cell NHL Stages 2-4 including the following nodal and extranodal subtypes:

Nodal:

* Peripheral T-cell lymphoma not otherwise specified (PTL NOS)
* Angioimmunoblastic lymphadenopathy (AILD)
* ALK 1 negative anaplastic large cell NHL

Extranodal:

* Hepatosplenic
* Enteropathy-associated
* Panniculitic

Exclusion Criteria:

* Previous treatment with chemotherapy or radiation with the exception of up to 1 cycle of CHOP chemotherapy.
* Expected survival < 4 months.
* ECOG performance status > 3.
* Inadequate haematologic function (Hb < 85g/L, ANC < 1000/mm3, or platelet count < 75,000/mm3) unless directly attributable to the NHL.
* Inadequate hepatic function (total bilirubin > 35μmol/L, alkaline phosphatase > 2x UL normal, AST/ALT > 2x UL normal)
* Inadequate renal function (serum creatinine > 130μmol/L), unless directly attributable to the NHL.
* Non-measurable or non-evaluable disease, according to criteria of Cheson et al49.
* Geographically inaccessible for follow-up
* Known hypersensitivity to study drugs
* Serious illnesses that may interfere with subject compliance, determination of causality of adverse events or would compromise other protocol objectives.
* Known HIV positivity or other pre-existing immunodeficiency (e.g., post-organ transplant).
* Known CNS involvement with lymphoma (tests to investigate CNS involvement are required only if clinically indicated).
* Pregnant or lactating women.
* Women who are of childbearing potential but are not using effective contraception. Men with reproductive potential who are not using effective contraception.
* Previous malignancy within the last 5 years with the exception of cervical carcinoma in situ or non melanoma skin cancer.
* Nasal natural killer (NK) T-cell NHL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2006-09; Primary Completion 2013-06 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
toxicity | 8 cycles of treatment

SECONDARY OUTCOMES:
efficacy | Post cycle 3 and Post cycle 8
tumour response | Post Cycle 3 and Post Cycle 8 Q 6 months in Followup
pharmacokinetic analysis | Day 1 of 8 Cycles of treatment and Post Last Dose on Day 3,6,10,13
immunological monitoring | Baseline Day 1 On Treatment Day 1 Cycle 4 and Cycle 8 and 6 months Follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Rena Buckstein, MD, Principal Investigator — Sunnybrook Health Sciences Centre, Odette Cancer Centre
Locations (5):
- Canada (5):
  - St. Paul's Hospital, Vancouver, British Columbia
  - Juravinski Cancer Centre, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Health Sciences Centre, Odette Cancer Centre, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario